CLINICAL TRIAL: NCT00229346
Title: Fibromyalgia and Psychiatric Symptoms Among PMS and PMDD Patients
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-04-3457-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Assessing FM and psychiatric disorder in patients suffering from PMS or PMDD

ELIGIBILITY:
Inclusion Criteria:

* PMDD
* PMS
* Referral to gynecologist clinic without symptoms of PMS or PMDD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel